CLINICAL TRIAL: NCT04220827
Title: A Phase I Study of Intraperitoneal Paclitaxel in Patients With Gastric Adenocarcinoma and Carcinomatosis or Positive Cytology
Brief Title: Paclitaxel for the Treatment of Gastric or Gastroesophageal Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0784; NCI-2019-08320 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0784 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-01-06; First posted 2020-01-07 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Clinical Stage IV Gastric Cancer AJCC v8; Clinical Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IVA Gastric Cancer AJCC v8; Clinical Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IVB Gastric Cancer AJCC v8; Clinical Stage IVB Gastroesophageal Junction Adenocarcinoma AJCC v8; Metastatic Gastric Adenocarcinoma; Metastatic Gastroesophageal Junction Adenocarcinoma; Pathologic Stage IV Gastric Cancer AJCC v8; Pathologic Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IVB Gastroesophageal Junction Adenocarcinoma AJCC v8; Peritoneal Carcinomatosis; Postneoadjuvant Therapy Stage IV Gastric Cancer AJCC v8; Postneoadjuvant Therapy Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVB Gastroesophageal Junction Adenocarcinoma AJCC v8
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (paclitaxel) (Experimental): Patients receive paclitaxel IP over 1 hour once weekly during weeks 1-3 and 5-7 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Given IP
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat

SUMMARY:
This phase I trial studies the side effects and best dose of paclitaxel for the treatment of gastric or gastroesophageal cancer. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the maximum tolerated dose (MTD) of paclitaxel via intraperitoneal route in subjects with gastric or gastroesophageal cancer and positive cytology or carcinomatosis.

SECONDARY OBJECTIVES:

I. Safety and tolerability of escalating doses of intraperitoneal paclitaxel in subjects with gastric or gastroesophageal cancer and positive cytology or carcinomatosis.

II. To make a preliminary assessment of the anti-tumor activity of paclitaxel in subjects with stage IV gastric or gastroesophageal cancer and positive cytology or carcinomatosis.

OUTLINE: This is a dose-escalation study.

Patients receive paclitaxel intraperitoneally (IP) over 1 hour once weekly during weeks 1-3 and 5-7 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Cytologic or histologic proof of adenocarcinoma of the stomach or gastroesophageal junction
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 60,000/Ul
* Serum creatinine =< 1.5 mg/dL
* Distant metastatic disease of peritoneum:

  * Positive peritoneal cytology
  * Carcinomatosis on diagnostic laparoscopy or laparotomy
  * Completion of preoperative systemic chemotherapy

Exclusion Criteria:

* Infections such as pneumonia or wound infections that would preclude protocol therapy
* Women with a positive urine or serum pregnancy test are excluded from this study; women of childbearing potential (defined as those who are not postmenopausal defined as no menses in greater than or equal to 12 months, have not had a hysterectomy or bilateral salpingo-ophorectomy, do not have ovarian failure, or have not had a surgical sterilization procedure) must agree to refrain from breast-feeding and practice adequate contraception as specified in the informed consent. Adequate contraception consists of oral contraceptive, implantable contraceptives, injectable contraceptives, a double barrier method, or abstinence. Men with reproductive potential must agree to an appropriate method of birth control, including abstinence or double barrier method (diaphragm plus condom)
* Subjects with unstable angina or New York Heart Association Grade II or greater congestive heart failure
* Subjects deemed unable to comply with study and/or follow-up procedures
* Subjects with a known hypersensitivity to protocol systemic chemotherapy that was life-threatening, required hospitalization or prolongation of existing hospitalization, or resulted in persistent or significant disability or incapacity
* Previous surgery that would preclude safe diagnostic laparoscopy with port placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to after 30 days after treatment completion
  Graded according to the National Cancer Institute Common Terminology Criteria for Adverse Safety data will be summarized using frequency tables by grade and attribution.

CONTACTS AND LOCATIONS:
Overall Officials: Brian D Badgwell, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/27/NCT04220827/ICF_000.pdf